CLINICAL TRIAL: NCT03824587
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy of Tenapanor as Adjunctive Therapy to Phosphate Binder Therapy in End-Stage Renal Disease (ESRD) Subjects With Hyperphosphatemia
Brief Title: Study to Evaluate the Efficacy of Tenapanor as Adjunctive Therapy to Phosphate Binder Therapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ardelyx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TEN-02-202
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Results first posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Hyperphosphatemia
MeSH Terms: conditions — Hyperphosphatemia | interventions — tenapanor; Sevelamer; ferric citrate; Calcium Carbonate; calcium acetate; sucroferric oxyhydroxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tenapanor 30 mg BID (Experimental): During the Double-Blind Treatment Period, subjects will receive tenapanor starting at a dose of 30 mg bid (three 10 mg tablets each time).
  Investigators may decrease or increase the dose of study medication based on s-P levels and/or gastrointestinal (GI) tolerability in 10 mg increments to a minimum of 10 mg bid or a maximum of 30 mg bid at any time during the Double-Blind Treatment Period.
  Interventions: Drug: Tenapanor; Drug: Phosphate Binder Agents
- Placebo (Placebo Comparator): same size, weight and appearance of experimental drug
  Interventions: Drug: Placebo; Drug: Phosphate Binder Agents

INTERVENTIONS:
Drug: Tenapanor — Active Drug
  Arms: Tenapanor 30 mg BID
Drug: Placebo — Inactive Drug
  Arms: Placebo
Drug: Phosphate Binder Agents — standard of care phosphate binder use at study entry was maintained throughout the entire study
  Other Names: sevelamer carbonate; ferric citrate; calcium carbonate; calcium acetate; sucroferric oxyhydroxide

SUMMARY:
This is a randomized, double-blind, placebo-controlled study to evaluate the effect of tenapanor on change in s-P levels when tenapanor is administered orally, twice daily for 28 days as adjunctive therapy to ESRD subjects with hyperphosphatemia on stable phosphate binder therapy.

DETAILED DESCRIPTION:
The study consists of a Screening visit; a Run-in Period of at least 2 weeks and up to 4 weeks, where existing phosphate binder treatment is maintained; and a 4-week Double-Blind Treatment Period.

At Screening, a subject must be on thrice daily phosphate binder therapy and have a serum phosphate (s-P) level ≥5.5 and ≤10.0 mg/dL to qualify for entering the study. s-P will be measured at each visit during the run-in period to enable the evaluation of the s-P randomization criteria.

Subjects who qualify to enroll in the study will be randomized in a 1:1 ratio to receive tenapanor or placebo while continuing their existing phosphate binder treatment.

During the Double-Blind Treatment Period, subjects will receive tenapanor or placebo starting at a dose of 30 mg bid

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent prior to any study specific procedures.
* Males or females aged 18 to 80 years, inclusive, at Screening
* Females must be non-pregnant, non-lactating and either be post-menopausal for at least -2 months, have documentation of irreversible surgical sterilization, use of acceptable -contraceptive method, or sexual abstinence, or a sterile sexual partner from Screening -until 30 days after the last subject visit.
* Males must agree to avoid fathering a child (or donating sperm), and therefore be either sterile (documented) or agree to use approved methods of contraception, from the time of enrollment until 30 days after end of study.
* Chronic maintenance hemodialysis (HD) 3x/week for at least 3 months or chronic maintenance peritoneal dialysis (PD) for a minimum of 6 months.
* If receiving active vitamin D or calcimimetics, the dose should have been unchanged for the last 4 weeks prior to Screening.
* Kt/V ≥1.2 at most recent measurement prior to Screening.
* Prescribed and taking phosphate binder medication at least 3 times per day, and the prescribed dose should have been unchanged during the last 4 weeks prior to Screening.
* Serum phosphorus levels must be ≥5.5 and ≤10.0 mg/dL at Screening and the end of the run-in period, analyzed at the central laboratory used in the study.

Exclusion Criteria:

* Severe hyperphosphatemia defined as having an s-P level >10.0 mg/dL on phosphate-binders at any time point during routine clinical monitoring for the 3 preceding months before Screening.
* Serum/plasma parathyroid hormone >1200 pg/mL.
* Clinical signs of hypovolemia at Screening as judged by the Investigator.
* History of inflammatory bowel disease (IBD) or irritable bowel syndrome with diarrhea (IBS-D).
* Scheduled for living donor kidney transplant or plans to relocate to another center during the study period.
* Use of an investigational agent within 30 days prior to Screening.
* Involvement in the planning and/or conduct of the study (applies to both Ardelyx/Contract Research Organization (CRO) staff and/or staff at the study site).
* If, in the opinion of the Investigator, the subject is unable or unwilling to fulfill the requirements of the protocol or has a condition which would render the results uninterpretable.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David P Rosenbaum, PhD, Study Chair — Ardelyx
Locations (48):
- United States (48):
  - Nephrology Consultants, LLC, Huntsville, Alabama
  - US Renal Care Pine Bluff, Pine Bluff, Arkansas
  - Southeast Renal Research, Beverly Hills, California
  - California Institute of Renal Research - Chula Vista, Chula Vista, California
  - North America Research Institute, Lynwood, California
  - DaVita Clinical Research - Santa Fe Spring, Montebello, California
  - Central Coast Nephrology, Salinas, California
  - North America Research Institute - San Dimas, San Dimas, California
  - Chabot Nephrology Medical Group, Union City, California
  - American Institute of Research, Whittier, California
  - Nova Clinical Research, LLC, Bradenton, Florida
  - Horizon Research Group - Coral Gables, Coral Gables, Florida
  - South Florida Research Institute, Lauderdale Lakes, Florida
  - Total Research Group, LLC, Miami, Florida
  - Omega Research Consultants, LLC, Orlando, Florida
  - Genesis Clinical Trials, Tampa, Florida
  - Dialysis Clinic, Inc - Albany GA, Albany, Georgia
  - Boise Kidney & Hypertension, PLLC - Meridian, Caldwell, Idaho
  - Renal Associates of Baton Rouge, Baton Rouge, Louisiana
  - Dialysis Clinic, Inc - Boston/Somerville, Boston, Massachusetts
  - Paragon Health PC - Nephrology Center, Kalamazoo, Michigan
  - InterMed Consultants, Minneapolis, Minnesota
  - Nephrology and Hypertension Associates, LTD, Tupelo, Mississippi
  - Clinical Research Consultants, LLC, Kansas City, Missouri
  - Dialysis Clinic, Inc - Kansas City, Kansas City, Missouri
  - Polack Renal, LLC (SMO), St Louis, Missouri
  - Kidney Specialists of Southern Nevada, Las Vegas, Nevada
  - Sierra Nevada Nephrology Consultants, Reno, Nevada
  - Dialysis Clinic, Inc - North Brunswick, North Brunswick, New Jersey
  - Renal Medicine Associates, Albuquerque, New Mexico
  - U.S. Renal Care - Gallup, Gallup, New Mexico
  - Northwell Health, Great Neck, New York
  - Mountain Kidney and Hypertension Associates, Asheville, North Carolina
  - Mountain Kidney & Hypertension Associates, P.A., Asheville, North Carolina
  - Durham Nephrology Associates, Durham, North Carolina
  - Southeastern Nephrology Associates - Wilmington, Wilmington, North Carolina
  - University of Cincinnati (UC) - Department of Nephrology, Cincinnati, Ohio
  - Northeast Clinical Research Center, Bethlehem, Pennsylvania
  - Columbia Nephrology Associates, P.A., Columbia, South Carolina
  - South Carolina Nephrology & Hypertension Center Inc., Orangeburg, South Carolina
  - DCI - Spartanburg, Spartanburg, South Carolina
  - Knoxville Kidney Center, PLLC, Knoxville, Tennessee
  - Med Center Dialysis, Houston, Texas
  - US Renal Care - Waxahachie, Mansfield, Texas
  - US Renal Care - Mesquite, Mesquite, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas
  - US Renal Care - Pleasanton Road, San Antonio, Texas
  - US Renal Care - Westover Hills, San Antonio, Texas

REFERENCES:
- [Derived] Sprague SM, Weiner DE, Tietjen DP, Pergola PE, Fishbane S, Block GA, Silva AL, Fadem SZ, Lynn RI, Fadda G, Pagliaro L, Zhao S, Edelstein S, Spiegel DM, Rosenbaum DP. Tenapanor as Therapy for Hyperphosphatemia in Maintenance Dialysis Patients: Results from the OPTIMIZE Study. Kidney360. 2024 May 1;5(5):732-742. doi: 10.34067/KID.0000000000000387. Epub 2024 Feb 7. PMID 38323855
- [Derived] Pergola PE, Rosenbaum DP, Yang Y, Chertow GM. A Randomized Trial of Tenapanor and Phosphate Binders as a Dual-Mechanism Treatment for Hyperphosphatemia in Patients on Maintenance Dialysis (AMPLIFY). J Am Soc Nephrol. 2021 Jun 1;32(6):1465-1473. doi: 10.1681/ASN.2020101398. Epub 2021 Mar 25. PMID 33766811

RESULTS

PARTICIPANT FLOW:
Groups:
- Tenapanor 30 mg BID: During the Double-Blind Treatment Period, subjects will receive tenapanor starting at a dose of 30 mg bid (three 10 mg tablets each time).
  Investigators may decrease or increase the dose of study medication based on s-P levels and/or gastrointestinal (GI) tolerability in 10 mg increments to a minimum of 10 mg bid or a maximum of 30 mg bid at any time during the Double-Blind Treatment Period.
  Tenapanor: Active Drug
  Phosphate Binder Agents: standard of care phosphate binder use at study entry was maintained throughout the entire study
Period: Run-in Period
Arm/Group | Tenapanor 30 mg BID | Placebo
Started | 0 (No subjects were on treatment during this period) | 511
Completed | 0 (No subjects were on treatment during this period) | 236
Not Completed | 0 | 275
Not completed — Screen Failure | 0 | 275
Period: Treatment Period
Arm/Group | Tenapanor 30 mg BID | Placebo
Started | 117 | 119
Completed | 112 | 116
Not Completed | 5 | 3
Not completed — Adverse Event | 4 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Kidney Transplant | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tenapanor 30 mg BID | Placebo | Total
Number analyzed (Participants) | 117 | 119 | 236
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.10 (12.326) | 53.88 (12.673) | 54.49 (12.491)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 45 | 97
  Male | 65 | 74 | 139
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 30 | 67
  Not Hispanic or Latino | 79 | 88 | 167
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 1 | 5
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 52 | 50 | 102
  White | 57 | 60 | 117
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Serum Phosphorus < 7.5 mg/dL [Count of Participants; unit: Participants] | 76 | 77 | 153
Serum Phosphorus >= 7.5 mg/d: [Count of Participants; unit: Participants] | 41 | 42 | 83
Sevelamer [Count of Participants; unit: Participants] | 57 | 58 | 115
Non-Sevelamer [Count of Participants; unit: Participants] | 60 | 61 | 121

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Phosphorus (s-P) Level From Baseline to Week 4.
Description: Difference in mean change from baseline in s-P level at Week 4 between the tenapanor and placebo groups.
Time Frame: 4 Weeks (28 days randomization period; from baseline to week 4)
Population: One patient did not receive study drug so was therefore not included in the modified ITT analysis
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Tenapanor 30 mg BID | Placebo
Number analyzed (Participants) | 116 | 119
mg/dL | -0.84 (0.131) | -0.19 (0.130)
Statistical Analysis 1: Comparison: Tenapanor 30 mg BID vs Placebo; Test type: Superiority; p = 0.0004, Mixed Models Analysis; Mean Difference (Net) = -0.65, 99% CI 2-sided [-1.13 to -0.18], Standard Error of Mean 0.182

2. Secondary Outcome: s-P Response at Week 4
Description: Achieving an s-P level <5.5 mg/dL
Time Frame: 4 Weeks (28 days randomization period)
Population: One patient did not receive study drug so was therefore not included in the modified ITT analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Tenapanor 30 mg BID | Placebo
Number analyzed (Participants) | 116 | 119
Participants | 43 | 26
Statistical Analysis 1: Comparison: Tenapanor 30 mg BID vs Placebo; Test type: Superiority; p = 0.0097, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.1

3. Secondary Outcome: Relative Change From Baseline in iFGF23 at Week 4
Description: iFGF23 at Week 4/baseline iFGF23 - 1
Time Frame: 4 Weeks (28 days randomization period)
Population: One patient did not receive study drug so was therefore not included in the modified ITT analysis
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Tenapanor 30 mg BID | Placebo
Number analyzed (Participants) | 116 | 119
pg/mL | 0.756 [0.686 to 0.834] | 0.931 [0.845 to 1.025]
Statistical Analysis 1: Comparison: Tenapanor 30 mg BID vs Placebo; Test type: Superiority; p = 0.0027, ANOVA

4. Secondary Outcome: Relative Change From Baseline in cFGF23 at Week 4
Description: cFGF23 at Week 4/baseline cFGF23 - 1
Time Frame: 4 Weeks (28 days randomization period)
Population: One patient did not receive study drug so was therefore not included in the modified ITT analysis
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Tenapanor 30 mg BID | Placebo
Number analyzed (Participants) | 115 | 119
pg/mL | 0.779 [0.716 to 0.848] | 0.947 [0.871 to 1.030]
Statistical Analysis 1: Comparison: Tenapanor 30 mg BID vs Placebo; Test type: Superiority; p = 0.0011, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the 4 week (28 days) treatment period.
Description: Adverse events were NOT collected during the run-in period since patients were receiving standard of care; any changes to health status during bhis period were reported in the medical history prior to randomization.
  The safety analysis includes all patients randomized (whether they received study drug or not).
Arm/Group | Tenapanor 30 mg BID | Placebo
All-Cause Mortality (participants affected / at risk) | 0/117 | 0/119
Serious Adverse Events (participants affected / at risk) | 3/117 | 5/119
Other Adverse Events (participants affected / at risk) | 50/117 | 8/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tenapanor 30 mg BID (N=117) | Placebo (N=119)
Acute Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cardiorespiratory Arrest (Cardiac disorders) | 1 | 0
Nodal Arrhythmia (Cardiac disorders) | 0 | 1
Arteriovenous Fistula Aneurysm (Injury, poisoning and procedural complications) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tenapanor 30 mg BID (N=117) | Placebo (N=119)
Diarrhea (Gastrointestinal disorders) | 50 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/87/NCT03824587/Prot_SAP_000.pdf